CLINICAL TRIAL: NCT01547195
Title: Assessment of the Effects of Swimming in the Treatment of Patients With Fibromyalgia.
Brief Title: Effects of Swimming in the Treatment of Fibromyalgia
Acronym: ESTF
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Giovana Fernandes, EVALUATION OF THE EFFECTS OF SWIMMING IN THE TREATMENT OF PATIENTS WITH FIBROMYALGIA, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0360/10
Record Dates: First submitted 2012-02-21; First posted 2012-03-07 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; swimming
MeSH Terms: conditions — Fibromyalgia | interventions — Swimming; Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group-swimming (Experimental)
  Interventions: Procedure: swim training
- Control-walk (Active Comparator)
  Interventions: Procedure: Training walk

INTERVENTIONS:
Procedure: swim training — Swimming training will be conducted with the implementation of the freestyle. The training will be held a week with 3 X 50 minutes for a period of 12 weeks.
  Patients will be monitored by a frequency waterproof. When at the beginning of training are carried out five minutes of heating, followed by 40minutos swimming 5 minutes and cooling at the end of training.
  Other Names: Swimming.; Freestyle.
  Arms: Group-swimming
Procedure: Training walk — The control group will perform walking exercise outdoors, monitored by a frequency, with the heart rate at anaerobic threshold assessed by cardiopulmonary exercise test.
  The training of walking will last 50 minutes, three times per week for 12 weeks.
  At the beginning of training, there will be a heating time of 5 minutes, followed by LA walk in cooling for 40 minutes and 5 minutes.
  Other Names: Walk.
  Arms: Control-walk

SUMMARY:
The recent scientific evidence shows that FM patients improve exercise capacity, symptoms and quality of life with the holding of regular exercise, especially aerobic exercise. Swimming is an aerobic workout of low impact, but no study has evaluated the effect of this activity in patients with fibromyalgia.

Randomized controlled trial with blinded evaluator, which will be evaluated patients with fibromyalgia were divided into two groups.

The intervention group will hold an exercise program of swimming (freestyle) and the other considered the control group held a walking program.

DETAILED DESCRIPTION:
Fibromyalgia (FM) is a syndrome characterized by diffuse musculoskeletal pain and chronic, with points called "hot spots", specific, sensitive and painful on palpation. Objective: To evaluate the efficacy of swimming in reducing the generally pain and improve the quality of function, of life and exercise capacity in patients with fibromyalgia. Material and Methods: 82 patients will be screened, diagnosed with fibromyalgia, who can swim the front crawl. Will be selected at UNIFESP outpatient clinics and also through advertisement in a newspaper. One group held the swimming training and the other group (control) will walk training. The Participants perform exercises (swimming or running) three times a week for 50 minutes, for 12 weeks. The exercises will be held at the anaerobic threshold determined by cardiopulmonary exercise testing. Measuring instrument: Questionnaires VAS (visual analogue scale) for pain, FIQ (Fibromyalgia Impact Questionnaire) to assess the quality of life related to disease, and also the SF-36 (short form health survey), which assesses quality of life in general. Cardiopulmonary stress test to assess cardiorespiratory fitness to sit and stand up and test to assess functional capacity. All participants will conduct an initial evaluation, after 6 and 13 weeks of training.

ELIGIBILITY:
INCLUSION CRITERIA:

* Female patients with fibromyalgia according to the classification criteria of the American College of Rheumatology;
* Patients with degree of pain between 4 and 8 cm by VAS-visual analog scale;
* Patients who can swim the freestyle "(crawl)"; Patients with stable-medication for at least three months;
* All patients will have signing the consent form.

EXCLUSION CRITERIA:

* Patients with uncontrolled cardiac disease and / or unable to perform aerobic exercises;
* Patients with severe psychiatric disorders;
* Patients with uncontrolled diabetes mellitus;
* Patients who practice regular physical exercise for at least 3 months;
* Patients with skin diseases that contraindicate the use of swimming pool;
* Patients with inflammatory rheumatic diseases.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-01 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Diminishing of pain | 3 months
  _ Assess the effectiveness of the practice of swimming in reducing pain and improving quality of life in patients with FM.

SECONDARY OUTCOMES:
Improving quality of life | 3 months
  _ Assess the effectiveness of the practice of swimming in improved function and aerobic capacity in patients with FM.

CONTACTS AND LOCATIONS:
Overall Officials: Giovana Fernandes, Mestranda, Principal Investigator — Universidade Federal de São Paulo
Locations (2):
- Brazil (2):
  - Ambulatory at UNIFESP, São Paulo, São Paulo
  - Universidade Federal de São Paulo, São Paulo, São Paulo

REFERENCES:
- [Derived] Fernandes G, Jennings F, Nery Cabral MV, Pirozzi Buosi AL, Natour J. Swimming Improves Pain and Functional Capacity of Patients With Fibromyalgia: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2016 Aug;97(8):1269-75. doi: 10.1016/j.apmr.2016.01.026. Epub 2016 Feb 20. PMID 26903145